CLINICAL TRIAL: NCT03400436
Title: Development of a Total Nutrient Index
Status: Completed | Type: Observational
Sponsor: National Institute of Health and Nutrition (Other Government)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Regan Bailey, Associate Professor, Purdue University
Other Study IDs: NCIR01_1
Record Dates: First submitted 2017-11-02; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Diet Habit
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention in observational studies — No intervention in observational studies

SUMMARY:
Dietary supplements are an important contributor to overall nutrient exposures for a large proportion of the U.S. population. Currently no standardized method exists to measure their use and contribution to total nutrient intakes, substantially limiting the rigor and reproducibility of their measurement. The purpose of this proposed project is to develop a standardized, data-driven, and valid metric that can be to measure use of and nutrient exposures from dietary supplements for use in research, clinical, and monitoring settings.

DETAILED DESCRIPTION:
Diet is a modifiable exposure that can positively or negatively impact health. More than half of adults and one-third of children use dietary supplements that contain nutrients critical to human health. Currently no metric exists to measure overall total nutrient exposures from all sources. Without measuring the contribution of dietary supplements, exposure classification is incomplete both for nutrient inadequacy and nutrient excess. Our highly qualified team proposes to develop the first comprehensive total nutrient index using a data-driven strategy with the nationally-representative National Health and Nutrition Examination Survey (NHANES). Indexes and scores are the preferred metric for use in nutrition because this method provides a standardized framework to compare across studies. In fact, the 2015 Dietary Guidelines for Americans Advisory Committee report, building on systematic reviews from the USDA Nutrition Evidence Library, were able to conclude that only diet classified by indexes and scores were useful for informing nutrition policy. The synthesis of the data in report yielded strong and consistent evidence for dietary patterns classified by indexes and scores and cardiovascular disease and weight status, and moderate evidence for dietary patterns and type 2 diabetes. However, no index or score is available that accounts for nutrients derived from dietary supplements and medications. In Aim 1, the investigators will develop a usual intake model that captures habitual intakes from food, beverages, dietary supplements, and medication, mitigiating the measurement error to the extent possible with self-reported dietary intakes. In Aim 2, the investigators will characterize the patterns of nutrients intake using data reduction techniques to create the most salient items to include in the index. The patterns will be carefully examined with regard to biomarkers, health behaviors, and measures of bone and body composition to create a scoring algorithm for the total nutrient index. In Aim 3, the investigators will test the reliability and the validity of the total nutrient index. The purpose of the total nutrient index is to provide a tool that can be used for research, monitoring, and policy purposes. Improving measures of dietary exposure will improve our ability to show causal links to health, ultimately enabling successful intervention strategies, and the use of the NHANES data to develop the total nutrient index greatly enhances its external validity.

ELIGIBILITY:
Inclusion Criteria:

* Children (</=18 years) and adults (>/=19 years) will be examined separately given the differential usage patterns in frequency and type of dietary supplements.

Exclusion Criteria:

* Pregnant and lactating females will be excluded from analysis because they are more likely to use dietary supplements than the general population.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NHANES is a nationally representative, cross-sectional continuous survey that includes non-institutionalized, civilian U.S. residents using a complex, stratified, multistage probability cluster sampling design. The NHANES data are publicly available and are released in 2-year datasets to ensure confidentiality of the participants and to allow for adequate sample size for statistical analysis. The NHANES data are planned and collected by the National Center for Health Statistics of the Centers for Disease Control and Prevention. Written informed consent is obtained for all participants or proxies and the survey protocol is approved by the research ethics review board at the National Center for Health Statistics. Currently, we plan to use NHANES 2011-2012 and 2013-2014 data cycles because these are the first to include oversampling of non-Hispanic Asian Americans and have supplement intake data collected on both the 24HRs and the 30-day frequency questionnaire.
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Nutrient quality index | NHANES 2011 to 2014
  This study will develop the nutrient quality index; this will be the tool used to measure nutrient quality in other studies.

IPD SHARING:
Plan to Share IPD: No
NHANES data are publicly available

REFERENCES:
- [Derived] Jun S, Cowan AE, Dodd KW, Tooze JA, Gahche JJ, Eicher-Miller HA, Guenther PM, Dwyer JT, Potischman N, Bhadra A, Forman MR, Bailey RL. Association of food insecurity with dietary intakes and nutritional biomarkers among US children, National Health and Nutrition Examination Survey (NHANES) 2011-2016. Am J Clin Nutr. 2021 Sep 1;114(3):1059-1069. doi: 10.1093/ajcn/nqab113. PMID 33964856
- [Derived] Cowan AE, Jun S, Tooze JA, Dodd KW, Gahche JJ, Eicher-Miller HA, Guenther PM, Dwyer JT, Moshfegh AJ, Rhodes DG, Bhadra A, Bailey RL. Comparison of 4 Methods to Assess the Prevalence of Use and Estimates of Nutrient Intakes from Dietary Supplements among US Adults. J Nutr. 2020 Apr 1;150(4):884-893. doi: 10.1093/jn/nxz306. PMID 31851315
- [Derived] Bailey RL, Dodd KW, Gahche JJ, Dwyer JT, Cowan AE, Jun S, Eicher-Miller HA, Guenther PM, Bhadra A, Thomas PR, Potischman N, Carroll RJ, Tooze JA. Best Practices for Dietary Supplement Assessment and Estimation of Total Usual Nutrient Intakes in Population-Level Research and Monitoring. J Nutr. 2019 Feb 1;149(2):181-197. doi: 10.1093/jn/nxy264. PMID 30753685